CLINICAL TRIAL: NCT06826053
Title: The Effect of Therapeutic Positions and the Smell of Breast Milk on Comfort and Vital Signs in Term Neonates With Respiratory Distress
Brief Title: The Smell of Breast Milk and Therapeutic Positions in Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Ayse Sonay Turkmen, Prof.Dr, Clinical Professor., Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: smell of breast milk
Record Dates: First submitted 2024-08-08; First posted 2025-02-13 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Distress
Keywords: respiratory distress; therapeutic position; the smell of breast milk; term neonatal
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic position group (Experimental): Therapeutic group
  Interventions: Other: Therapeutic position
- Therapeutic position + smell of breast milk (Experimental): Therapeutic position + smell of breast milk
  Interventions: Other: Therapeutic position + smell breast milk

INTERVENTIONS:
Other: Therapeutic position — each newborn was given four different therapeutic positions in sequence.
  Arms: Therapeutic position group
Other: Therapeutic position + smell breast milk — each newborn will be given four different therapeutic positions in sequence and will be made to smell the scent of breast milk.
  Arms: Therapeutic position + smell of breast milk

SUMMARY:
Before starting the data collection process, a pilot study was conducted with 10 preterm newborns, five in the safe swaddling group and five in the control group, to evaluate the comprehensibility of the questionnaire form and the feasibility of the application. The newborns included in the pilot study were not included in the study.

At the beginning of the study, parents of newborns who met the sample selection criteria were informed about the purpose and content of the study and informed consent was obtained from those who agreed to participate in the study. Data were obtained from parents of infants 38 weeks and older who were hospitalized in the Tertiary NICU and who met the sample selection criteria by using data collection tools. Firstly, parents were informed about the study through the "Information and Informed Consent Form" (Appendix-E). They were included in the study if they volunteered. Written informed consent was obtained from the parents who volunteered to participate in the study. Data were collected using "Data Collection Tools" prepared by the researcher.

Newborns will be randomly divided into two groups;

* Group 1: Therapeutic position
* Group 2: Therapeutic position + the smell of breast milk Number, percentage, mean and standard deviation will be used in the descriptive statistics of the study. The normality of the data will be evaluated with the Kolmogrow Smirnow test. Kappa analysis will be used in the evaluation of inter-observer agreement. Chi-square test will be used for the comparison of categorical data, t test and Anova in independent groups will be used for the comparison of normally distributed data, Friedman, Wilcoxon, Mann Whitney U and Kruskal Wallis tests will be used for the comparison of non-normally distributed data. Within-group evaluation will be evaluated by repeated measures analysis of variance. Significance level p<0.05 will be accepted.

Continuous data will be shown as mean ± standard deviation for normally distributed data, median and 25-75th quartile for non-normally distributed data, and frequency and percentage for categorical data. For comparisons of differences between categorical variables by groups, Pearson chi-square test will be used for RxC tables with expected observations of 5 and above and Fisher Freeman Halton test will be used for RxC tables with expected observations below 5.

DETAILED DESCRIPTION:
Ethical and institutional permissions were obtained before starting to collect the data. Written consent will be obtained from all parents via a voluntary consent form. Newborns will be randomly selected into 2 groups.

Group 1: term neonates in four different therapeutic positions (prone-right lateral-supine-left lateral). The positions of the newborns will be changed every two hours in sequence. In addition, peak heart rate, respiration, oxygen saturation, comfort (2 observers), pain (2 observers), distress (2 observers) will be evaluated every 30 minutes for two hours. A total of 5 measurements and evaluations will be performed.

Group 2: Therapeutic position + the smell of breast milk . The positions of the newborns will be changed every two hours in sequence. Newborns in this group will also be made to smell the odor of breast milk. For breast milk odor, approximately 3-5 cc of breast milk obtained from each baby's own mother's milk will be dripped onto 4x4 gauze swabs. These gauze pads dripped with breast milk will be placed at a distance of approximately 10 cm from the baby's nose. Then, peak heart rate, respiration, oxygen saturation, comfort (2 observers), pain (2 observers), distress (2 observers) values of the newborn will be evaluated every 30 minutes for two hours. A total of 5 measurements and evaluations will be performed.

Hypotheses of the Study H1: Different therapeutic positions given to newborns have an effect on respiratory rate.

H2: Different therapeutic positions given to newborns have an effect on peak heart rate.

H3: Different therapeutic positions given to newborns have an effect on oxygen saturation.

H4: Different therapeutic positions given to newborns have an effect on comfort level.

H5: Different positions given to newborns and breast milk odor have an effect on respiratory rate.

H6: Different positions given to newborns and breast milk odor have an effect on peak heart rate.

H7: Different positions given to newborns and breast milk odor have an effect on oxygen saturation.

H8: Different positions given to newborns and breast milk odor have an effect on comfort level.

H9: There is a significant difference between the two groups in terms of respiratory rate of newborns.

H10: There is a significant difference between the two groups in terms of peak heart rate of newborns.

H11: There is a significant difference between the two groups in terms of oxygen saturation of newborns.

H12: There is a significant difference between the two groups in terms of comfort level of newborns.

ELIGIBILITY:
Inclusion Criteria:

* NICU admission immediately after birth.
* The babies were term births (births at 38 weeks and above).
* The baby was not given analgesics and/or sedatives.
* The baby had spontaneous breathing.
* Families' acceptance to participate in the study.

Exclusion Criteria:

* With a thoracic tube, umbilical vein catheter or dialysis catheter.
* With active infection.
* Tachypnea and unstable oxygen saturation ≤ 90%.
* Receiving sedation therapy.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
heart rate | every 30 minutes for two hours
  heart rate
oxygen saturation values | every 30 minutes for two hour
  oxygen saturation values
respiratory rate | every 30 minutes for two hours
  respiratory rate

SECONDARY OUTCOMES:
Neonatal Comfort Behavior Scale Score | every 30 minutes for two hours
  comfort scale

CONTACTS AND LOCATIONS:
Locations (1):
- Karamanoglu Mehmetbey University, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No